CLINICAL TRIAL: NCT04264026
Title: Open-label Phase 2 Study of MDMA-Assisted Psychotherapy in Veterans With Combat-Related, Refractory PTSD
Brief Title: MDMA-Assisted Psychotherapy in Veterans With Combat-Related, Refractory PTSD
Acronym: VALLMDMA_001
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: VA Loma Linda Health Care System (U.S. Federal Agency)
Collaborators: Multidisciplinary Association for Psychedelic Studies (Other)
Responsible Party: Principal Investigator, Shannon Remick, Principal Investigator, VA Loma Linda Health Care System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1311
Record Dates: First submitted 2020-02-07; First posted 2020-02-11 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Post Traumatic Stress Disorder; Combat Stress Disorders
Keywords: Veterans; Refractory PTSD; PTSD; MDMA
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Combat Disorders | interventions — N-Methyl-3,4-methylenedioxyamphetamine

STUDY DESIGN:
Intervention Model Description: Single-site, open-label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open Label (Experimental): Participants will receive an initial dose of 80 mg of 3,4-methylenedioxymethamphetamine (MDMA) and an optional supplemental dose of 40 mg MDMA during the first Experimental Session. In the second and third Experimental Sessions, the participant will receive an initial dose of 120 mg MDMA and an optional supplemental dose of 40 mg MDMA.
  Interventions: Drug: 3,4-methylenedioxymethamphetamine

INTERVENTIONS:
Drug: 3,4-methylenedioxymethamphetamine — Bottles are labeled with a unique container number, protocol number, IMP name, lot number, sponsor name and a statement that the IMP is restricted to clinical trial use only.
  Other Names: MDMA

SUMMARY:
This will be a single-site, open-label phase 2 study designed to test the feasibility of administering MDMA in conjunction with psychotherapy for combat-related treatment-resistant PTSD in US military veterans currently enrolled in VA. MDMA will be given in conjunction with structured psychotherapy in three single-dose psychotherapy sessions in a hospital setting over the course of 12 weeks, along with preparatory and integration psychotherapy sessions in-between each active-dose session. The overall objective of this study is to evaluate the risks, benefits, and feasibility of MDMA used in conjunction with manualized psychotherapy, on reduction of symptoms, or remission of PTSD, as evaluated by standard clinical measures, in a VA Healthcare System.

The primary outcome measure for the study is the Clinician-Administered PTSD Scale (CAPS-5), a semi-structured interview used in the majority of clinical trials for PTSD, which will be assessed at baseline, primary endpoint, and at the long-term 12-month follow-up visit. Secondary safety and efficacy measures will also be collected.

The planned duration of this study is 1-3 years, with each active treatment period lasting approximately 12 weeks, along with a long-term follow-up 12 months after the last active-drug session.

DETAILED DESCRIPTION:
This will be a single-site, open-label study, investigating the use of MDMA-assisted psychotherapy for treatment-resistant combat-related PTSD. This study will consent up to 50 current-era combat veterans for study and the first 10 participants who meet criteria will be eligible to receive study medication. Any patient who drops out before the third Experimental Session will be replaced. Dropout rates will be recorded. In this protocol, enrollment is defined as the time the participant signs informed consent. Time from initial screening/enrollment to collection of the primary endpoint will last approximately 12-18 weeks. To assess durability of treatment, participants will be assessed approximately 12 months after the last MDMA session for the long-term follow-up. The study will consist of a prescreening/screening/enrollment period, three pre-experimental (preparatory) dose psychotherapy sessions (spaced approximately one week apart), three experimental dose therapy sessions, nine integrative follow-up sessions, one assessment of primary endpoint, and a long-term 12-month follow-up assessment. Psychiatric medication tapering will occur after eligibility confirmation (after completion of baseline CAPS-5, prior to Experiential Sessions) to allow for appropriate medication washout.

The primary objective of this study is to evaluate the safety and effectiveness of MDMA in Veterans with combat-related, refractory PTSD when used in conjunction with manualized psychotherapy on reduction of symptoms, or remission of PTSD, as evaluated by standard clinical measures.

Effectiveness will be measured by evaluating the change in CAPS-5 scores from baseline to the primary endpoint. Primary endpoint will be collected 2 months after the third Experimental Session with MDMA. To access long-term effectiveness, CAPS-5 will also be collected at the long-term follow-up.

Secondary Objectives:

1. Assess changes in self-reported PTSD symptoms as measured with the PTSD-symptom checklist at screening and baseline, during most face-to-face visits, at the primary endpoint, and during the long-term follow-up.

   a. Life Event Checklist (LEC) for PCL-5 will be administered at baseline (screening), primary endpoint, and long-term follow-up.
2. Assess depression symptoms with the Beck Depression Inventory-II (BDI-II) at baseline (screening), primary endpoint, and long-term 12-month follow-up.
3. Assess changes in alcohol consumption.

   1. The AUDIT-C (Alcohol Use Disorders Identification Test) will be used to measure baseline alcohol use over the past year prior to study entry (at screening) and at long-term follow up.
   2. Alcohol use starting after study screening will be monitored based on participants self-report. Participants will be directed to keep a Drinking Diary throughout the study measuring the number of standard alcoholic beverages consumed per day. Drinking Diary for each participant will be collected weekly until their last psychotherapy visit. Participants will continue to record weekly alcohol use on their own until collection at the primary endpoint.
4. Assess changes in drug consumption.

   a. Drug Use Disorders Identification Test (DUDIT) will be assessed at baseline (screening) and at long-term follow-up).
5. Assess changes in self-reported sleep quality via the Pittsburgh Sleep Quality Index (PSQI) from baseline (screening) to primary endpoint and long-term 12-month follow-up.
6. Assess changes in posttraumatic growth via Post Traumatic Growth Inventory (PTGI) scores from baseline (at screening) to primary endpoint and long-term 12-month follow-up.
7. Healthcare utilization will also be assessed by retrospective chart review.

Twelve months after the final Experimental Session, the long-term effects of MDMA-assisted psychotherapy on symptoms of PTSD will be assessed via CAPS-5 and PCL-5 with LEC, alcohol use via AUDIT, drug use behaviors via DUDIT, depression via BDI-II, self-reported sleep quality via PSQI, post-traumatic growth via PTGI, suicidality via C-SSRS, and response to research participation via RRPQ (Reactions to Research Participation Questionnaire).

Participants will also be assessed for suicidality at every face-to-face visit.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be eligible for VA healthcare and currently being treated by VA Loma Linda Healthcare System or VA Long Beach providers
2. Participants must meet DSM 5 criteria for combat-related PTSD (within the past 6 months). PTSD must be defined as treatment-resistant.
3. Participants must have been exposed to combat in the current-era war.
4. Participants must be 18-55 years old.
5. Participants must be generally healthy overall without any significant medical comorbidities (see exclusion criteria).
6. Participants must be willing to refrain from alcohol for 72 hours prior to each MDMA session and be deemed not at risk for significant alcohol withdrawal.
7. Participants must be willing to refrain from taking any psychiatric medications during the study period, including gabapentin or any other anticonvulsants. If they are being treated with psychoactive medications during recruitment, participants must be willing and determined safe (by study physician(s)) to undergo medically-supervised withdrawal from these medications. The medications will be withdrawn in an appropriate fashion to minimize any withdrawal effects. The participants must be able to refrain from starting any new medications during the study period. The only exception to this will be in the case of rescue medications that may be administered in the event of a crisis during the experimental study sessions.
8. Agree that, for one week preceding an MDMA session will refrain from:

   1. Taking any herbal supplement (except with prior approval of the research team);
   2. Taking any nonprescription medications (with the exception of non-steroidal anti-inflammatory drugs or acetaminophen unless with prior approval of the research team);
   3. Taking any prescription medications, with the exception of birth control pills, thyroid hormones or other medications approved by the research team.
9. Are proficient in speaking and reading English.
10. Must meet capacity and consent for treatment.
11. Participants who are engaged in non-PTSD psychotherapy at the time of study screening, may continue to see their therapist during the course of the study. If seeing a non-VA therapist, participants must sign a release for the investigators to communicate directly with their therapist. Subjects may not change therapists, increase the frequency of therapy or commence any new type of therapy until after the evaluation session 2 months after the final experimental session.
12. Participants of childbearing potential and age must have a negative pregnancy test and must agree to use an effective form of birth control during the study period.
13. Participants must be willing to stay overnight at the hospital after each experimental session.
14. Agree to have transportation other than driving themselves home on the day after an MDMA session.
15. Are willing to follow restrictions and guidelines concerning medications, consumption of food, beverages, alcohol, nicotine, or illicit substances.
16. Must provide a contact (relative, spouse, close friend or other caregiver) who is willing and able to be reached by the investigators in the event of a participant becoming suicidal.
17. Must agree to inform the investigators within 48 hours of any medical conditions and procedures.
18. Agree to not participate in any other interventional clinical trials during the duration of this study.
19. Must be able to swallow pills.

Exclusion Criteria:

1. Individuals with only non-combat related PTSD. Note: participants will not be excluded for having multiple traumas so long as one of those is combat-related.
2. Participants currently engaged in PTSD psychotherapy.
3. Individuals that are determined medically unstable, unsafe for outpatient detoxification from alcohol, at risk for severe alcohol withdrawal, or unwilling/unable to refrain from alcohol use for at least 72 hours prior to experimental session.
4. Lack a stable living situation or supportive system.
5. Any person unable to give adequate informed consent.
6. Participants of childbearing potential who are pregnant, nursing, or of childbearing age unwilling/unable to practice an effective means of birth control.
7. People with a history of, or a current psychotic disorder, dissociative disorder, bipolar affective disorder or personality disorders.
8. Have a current eating disorder.
9. Have current major depressive disorder with psychotic features.
10. Would present a serious risk to others as established through clinical interview and contact with treating psychiatrist.
11. People with evidence or history of significant hematological, cardiovascular, cerebrovascular, coronary, pulmonary, endocrine, renal, gastrointestinal, hepatic (including LFTs > 3x upper limit of normal), immunocompromising (examples include recent organ transplant and required to be on immunosuppressants, those with HIV/AIDs, cancer or an autoimmune disease [i.e., lupus, multiple sclerosis, rheumatoid arthritis]), neurological disease (including seizure disorder or cognitive impairment). Patients with hypothyroidism who are on adequate and stable thyroid replacement will not be excluded.
12. Have uncontrolled hypertension using the standard criteria of the American Heart Association (values of 140/90 milligrams of Mercury [mmHg] or higher assessed on three separate occasions).
13. Have a marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval >450 milliseconds [ms] for men or >470 ms for women corrected by Bazett's formula).
14. Have a history of additional risk factors for Torsade de pointes (e.g., heart failure, hypokalemia, family history of Long QT Syndrome).
15. Require use of concomitant medications that prolong the QT/QTc interval during Experimental Sessions.
16. Have history of hyponatremia or hyperthermia.
17. People weighing less than 50 kg.
18. People with prior use of "Ecstasy" (illicit drug preparations purported to contain MDMA) more than ten times within the past ten years or at any time within the past 6 months or have previously participated in a MAPS-sponsored MDMA clinical trial.
19. People with ketamine use within the last 12 weeks.
20. People with a serious suicide risk or who are likely to require hospitalization within the course of the study.
21. Individuals who require ongoing treatment with psychoactive medications.
22. Individuals meeting DSM-5 criteria for active substance use disorder for any substance other than caffeine or nicotine assessed.
23. Patients in a residential or intensive outpatient treatment program for substance use will be excluded (patients engaged in self-help program such as after care and relapse prevention and alcoholics-anonymous can be included).
24. Have received Electroconvulsive Therapy (ECT) within 12 weeks of enrollment.
25. Currently engaged in compensation litigation whereby financial gain would be achieved from prolonged symptoms of PTSD or any other psychiatric disorders.
26. Unable to ensure reliable transportation to and from study visits or have unstable housing.
27. Any potential participant presenting current serious suicide risk, as determined through psychiatric interview, responses to questionnaires, and clinical judgment of the investigator will be excluded; however, history of suicide attempts is not an exclusion. Any participant who is likely to require hospitalization related to suicidal ideation and behavior will be excluded.
28. Any potential participant with a C-SSRS Suicidal Ideation score of 5 during the prior six months, or with a suicidal ideation of 4 occurring more frequently than one day per week within the past month will be excluded.
29. Regardless of C-SSRS score, any participant presenting current serious suicide risk, as determined through psychiatric interview, responses to C-SSRS, and clinical judgment of the investigator will be excluded; however, history of suicide attempt is not an exclusion. Any participant who is likely to require hospitalization related to suicidal ideation and behavior will be excluded.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2021-07-29 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Change in total score of CAPS-5 | baseline, primary outcome (2 months after last experimental/MDMA session), 12-month follow-up
  The primary objective was amended in January 2024. The study will now aim to explore the feasibility of MDMA used in conjunction with manualized psychotherapy on reduction of symptoms, or remission of combat-related treatment resistant PTSD, as evaluated by standard clinical measures as a multiple case series.

SECONDARY OUTCOMES:
Changes in self-reported PTSD symptoms | baseline, primary outcome (2 months after last experimental/MDMA session), 12-month follow up
  Assess changes in self-reported PTSD symptoms as measured with the PTSD-symptom checklist (PCL-5)
Depression Symptoms | through study completion, an average of 1 year
  Assess depression symptoms with the Beck Depression Inventory-II. The Beck Depression Inventory-II (BDI-II) is a 21-item self-report measure of depressive symptoms, with scores ranging from 0 to 63, higher scores indicative of greater (more severe) depression.
Changes in Alcohol Consumption | through study completion, an average of 1 year
  Assess changes in alcohol consumption.
  1. The AUDIT-C (Alcohol Use Disorders Identification Test) will be used to measure baseline alcohol use over the past year prior to study entry (at screening) and at long-term follow up (V18).
  2. Alcohol use starting after study screening will be monitored based on participants selfreport.
  Participants will be directed to keep a Drinking Diary throughout the study measuring the number of standard alcoholic beverages consumed per day.
Changes in Drug Consumption | Baseline (screening) and long-term 12-month follow up (V18)
  Drug Use Disorders Identification Test (DUDIT) will be assessed
Changes in self-reported sleep quality | through study completion, an average of 1 year
  Assess changes in self-reported sleep quality via the Pittsburgh Sleep Quality Index (PSQI). It consists of 19 items, with possible responses ranging from 0 to 4 on a five-point scale. Global scores can range from 0 to 21, with higher scores reflecting poorer sleep quality, and a score below 5 indicating good sleep.
Changes in posttraumatic growth | through study completion, an average of 1 year
  Assess changes in posttraumatic growth via Post Traumatic Growth Inventory (PTGI) scores. The Post Traumatic Growth Inventory (PTGI)115-116 is a 21-item self-report measure of perceived growth or benefits occurring after a traumatic event. It contains five subscales- relationship to others, new possibilities, personal strength, spiritual change, and appreciation of life. Higher scores implies that the person has undergone a positive transformation.
Healthcare Utilization | Baseline through study completion, an average of 1 year
  Healthcare utilization will also be assessed by retrospective chart review to determine psychotherapy treatment history in comparison from baseline to study end.

CONTACTS AND LOCATIONS:
Overall Officials: Shannon Remick, MD, Principal Investigator — Staff Psychiatrist
Locations (1):
- VA Loma Linda Health Care System, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No
No sharing planned

DOCUMENTS (1):
  • Informed Consent Form (2023-03-01): https://cdn.clinicaltrials.gov/large-docs/26/NCT04264026/ICF_000.pdf